CLINICAL TRIAL: NCT05578950
Title: Comparative Study Between Pulse Therapy With Oral Itraconazole Versus Continuous Oral Terbinafine Therapy for Treatment of Onychomycosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Dr Mahboob Ali, principal investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cmh abbottabod
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — Itraconazole; Terbinafine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A pulse therapy of itraconazole (Active Comparator): patients with pulse therapy group recieved oral itraconazole 100 mg, two capsules twice daily for 7 days a month
  Interventions: Drug: itraconazole
- group B continous therapy of terbinafine (Active Comparator): patients with continous therapy group , recieved continous oral 250 mg terbinafine once daily for 12 weeks continously
  Interventions: Drug: terbinafine

INTERVENTIONS:
Drug: itraconazole — 100 mg two capsules of itraconazole were givev twice daily to 50 patients in group A for one week per month . baseline LFTs were also monitered
  Other Names: capsules icon
  Arms: group A pulse therapy of itraconazole
Drug: terbinafine — one 250 mg tablet of terbinafine were given once daily to 50 patients in group B for 12 weeks continously
  Other Names: tablets terbesil
  Arms: group B continous therapy of terbinafine

SUMMARY:
Nail fungus, often known as onychomycosis (OM), can attack either the toenails or the fingernails. Onychomycosis can affect the matrix, the nail bed, or the nail plate. Though not fatal, onychomycosis is a significant condition that can impede a person's mobility and ability to work. Onychomycosis's wide-ranging emotional and social impacts can have a serious negative impact on patients' well-being.

White superficial onychomycosis (WSO), proximal subungual onychomycosis (PSO), endonyx onychomycosis (EO), and candidal onychomycosis are the most common subtypes of onychomycosis. A patient may exhibit characteristics from more than one of these categories. A severe case of onychomycosis, regardless of its subtype, is called total dystrophic onychomycosis.

Different types of onychomycosis have different pathophysiology. The most frequent type of onychomycosis, known as distal lateral subungual onychomycosis, occurs when a fungus travels from the plantar skin to the nail bed through the hyponychium.

These sections of the nail apparatus become inflamed, leading to the outward manifestations of distal lateral subungual onychomycosis. White superficial onychomycosis, on the other hand, is a less common presentation produced by invasion of the nail plate's surface. Fungi colonise the deep section of the proximal nail plate in the rare condition known as proximal subungual onychomycosis. When the fungi infect the nail through the skin and penetrate the nail plate, the result is known as endonyx onychomycosis, a subtype of distal lateral onychomycosis.

Over and over again, terbinafine has been shown to be more effective than other antifungal medicines in clinical trials. Mycological cure rates for onychomycosis were 76% with terbinafine, 63% with pulse itraconazole, and 48% with fluconazole, according to a meta-analysis of 18 studies.

The aim of this study is to determine the aim of this study is to compare pulse therapy with oral itraconazole versus continuous oral terbinafine for treatment of onychomycosis

ELIGIBILITY:
Inclusion Criteria:

* patients age between 18 and 60 years
* patients positive for fungus via direct microscopy due to identification of hyphae or blastospores on the toe nails
* patients having positive fungal culture
* patients who had not applied any topical agent to the target toe nail for the last one month

Exclusion Criteria:

* Pregnant patients
* Lactating women
* Patients with poor adherence
* Patients previously allergic to oral itraconazole or terbinafine
* Patients with elevated baseline LFTs such as ALT ,AST , alkaline phosphatase and total bilirubin twice the upper limit of normal
* History of renal disease
* Patients unresponsive to systemic antifungal therapy with in the past year
* History of using systemic immunosuppressants
* Immunocompromised patients
* Pateints with ventricular dysfunction and history of congestive heart failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
effectiveness of pulse therapy of itraconazole and continuous therapy of terbinafine for the treatment of onychomycosis as assessed by ONYCHOMYCOSIS SEVERITY INDEX (OSI) | 12 weeks
  OSI is calculated as follows:score of area involvement multiplied by score for proximity of disease to the matrix and10 points are added for the presence of dermatophytoma or subungal hyperkeratosis of greater than 2 mm.
  A cumulative score of 0 indicates cured; 1 through 5, mild onychomycosis; 6 through 15, moderate onychomycosis; and 16 through 35 , severe onychomycosis.
  Area of involvement score 0 to 5, proximity of disease to matrix score 1 to 5 , presence of subungal dermatophytoma or subungal hyperkeratosis score 0 or 10

CONTACTS AND LOCATIONS:
Locations (1):
- Cmh Abbottabad, Abbottābād, Khyber Pakhtunkhwa, Pakistan